CLINICAL TRIAL: NCT07106268
Title: Aqueous Humor Proteome Analysis in Conbercept-treated Retinal Vein Occlusion With Macular Edema
Brief Title: Aqueous Humor Proteome in Retinal Vein Occlusion With Macular Edema
Status: Active, not recruiting | Type: Observational
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Chuanzhen Zheng, Principal investigator, Tianjin Medical University Eye Hospital
Other Study IDs: MR-12-24-035937
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Aqueous humor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with central retinal vein occlusion: Received three injections of the anti-VEGF drug Conbercept
- Patients with branch retinal vein occlusion: Received three injections of the anti-VEGF drug Conbercept
- Cataract patients without other eye diseases and other chronic diseases: Undergo cataract surgery

SUMMARY:
the goal of this observational study is to the find the molecular mechanisms underlying the prognosis process of Retinal vein occlusion in patients with retinal vein occlusion . The main question it aims to answer is:

What are the changes in protein in the aqueous humor during treatment in patients who are sensitive to anti-VEGF drug therapy?

ELIGIBILITY:
Inclusion Criteria:

* Cystic or diffuse edema in the macular area, retinal vein tortuous dilation with hemorrhage
* Optical coherence tomography (OCT) examination showed that the macular area was raised, edema and thickened
* Monocular disease, baseline central retinal thickness (CRT) ≥ 250mm
* Intravitreal injection, laser photocoagulation and blood circulation and blood stasis removal drugs were not treated before surgery
* The patient had normal blood pressure, negative urine protein, normal liver and kidney function, and normal electrocardiogram

Exclusion Criteria:

* Patients with fluorescein fundus angiography (FFA) showing a large area (10 optic disc areas) without perfusion requiring retinal photocoagulation
* Patients with chronic dacryocystitis, glaucoma, cataract, severe proliferative vitreoretinopathy or vitreous hemorrhage, epi macular membrane or macular ischemia, diabetic retinopathy, age-related macular degeneration, ocular trauma and other diseases
* Intravitreal therapy or laser photocoagulation with corticosteroids or anti-VEGF drugs within three months before the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with retinal vein occlusion with macular edema
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Central retinal thickness | March 2023 - June 2024
  The Heidelberg Optical Coherence Tomography scanner was used to detect the central retinal thickness in patients

SECONDARY OUTCOMES:
Best corrected visual acuity | March 2023 - June 2024
  BCVA was measured using logarithm of the minimum angle of resolution (LogMAR) chart

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hospital, Tianjin, Province, China

IPD SHARING:
Plan to Share IPD: No